CLINICAL TRIAL: NCT04724694
Title: Brief Cognitive Behavioral Therapy for Chronic Pain to Improve Functional Outcomes Among Primary Care Veterans
Brief Title: Brief Cognitive Behavioral Therapy for Chronic Pain to Improve Functioning Among Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3485-R; RX003485-01A1 (Other Grant/Funding Number: VA-ORD)
Record Dates: First submitted 2021-01-14; First posted 2021-01-26 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Pain; Pain
Keywords: primary care; chronic pain; cognitive behavioral therapy; integrated primary care; musculoskeletal pain
MeSH Terms: conditions — Musculoskeletal Pain; Pain; Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two arm parallel design: 1) primary care treatment as usual, or 2) primary care treatment as usual and Brief Cognitive Behavioral Therapy for Chronic Pain
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief CBT for Chronic Pain and treatment as usual (Experimental): Participants will receive Brief CBT-CP in addition to usual primary care treatment. Brief CBT-CP is a manualized protocol that includes six, 30-minute sessions over the course of 6-12 weeks. Session one focuses on foundational pain education and the development of treatment goals. Session two emphasizes balanced engagement in physical activity and pleasurable events. Session three emphasizes skills training for easily implemented relaxation techniques. Sessions four and five focus on recognizing and modifying unhelpful thoughts that negatively impact pain. Session six focuses on relapse prevention and independent implementation of CBT-CP skills following treatment.
  Interventions: Behavioral: Brief CBT for Chronic Pain; Other: Treatment as usual
- Treatment as usual only (Other): Participants assigned to treatment as usual will receive standard medical care from their primary care provider including pain medications, brief advice (e.g., use of relative rest, application of heat or ice, other self-care strategies), or referral to pain-related adjunctive interventions (e.g., physical therapy), as indicated.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Brief CBT for Chronic Pain — Brief CBT-CP is a manualized protocol that includes six, 30-minute sessions over the course of 6-12 weeks. Session one focuses on foundational pain education and the development of treatment goals. Session two emphasizes balanced engagement in physical activity and pleasurable events. Session three emphasizes skills training for easily implemented relaxation techniques. Sessions four and five focus on recognizing and modifying unhelpful thoughts that negatively impact pain. Session six focuses on relapse prevention and independent implementation of CBT-CP skills following treatment.
  Other Names: Brief CBT-CP
  Arms: Brief CBT for Chronic Pain and treatment as usual
Other: Treatment as usual — Participants assigned to TAU will receive standard medical care from their primary care provider including pain medications, brief advice (e.g., use of relative rest, application of heat or ice, other self-care strategies), or referral to pain-related adjunctive interventions (e.g., physical therapy), as indicated.
  Other Names: Primary care treatment as usual

SUMMARY:
Chronic pain is very common among primary care Veterans and can seriously impact overall patient functioning and well-being. Currently, behavioral treatments for pain management are not often provided in primary care because they are designed to be delivered in specialty care settings, such as chronic pain clinics. To address this gap in care, the proposed study will test if Brief Cognitive Behavioral Therapy for Chronic Pain (Brief CBT-CP) is an effective treatment. Therefore, the first objective of the proposed study is to conduct a randomized controlled trial of Brief CBT-CP compared to primary care treatment as usual to assess treatment effectiveness by examining changes in pain-related physical activity interference, psychological distress, pain intensity, and other related outcomes. 178 eligible participants will be randomized into either Brief CBT-CP and primary care treatment as usual or primary care treatment as usual only. Eligible Veterans will include those with chronic musculoskeletal pain and pain-related functional impairment identified from primary care. Participants assigned to Brief CBT-CP will receive six sessions of treatment in 30-minute appointments. This intervention will include education and goal setting, activities and pacing, relaxation skills, cognitive coping, and relapse prevention. Assessments will include validated self-report measures that will take place at pre-treatment (baseline), mid-treatment, post-treatment, and at 6-month follow-up. The second objective of this study is examine the mechanisms by which Brief CBT-CP leads to improvement in patient outcomes. Statistical analysis will reveal if changes pain self-efficacy (i.e., perceived ability to manage pain or engage in usual activities despite being in pain) and catastrophizing (i.e., unhelpful, negative though patterns about pain and pain management) lead to improvements in patient functioning. The third objective of this study will be to explore perceptions of Brief CBT-CP among patients who experience significant improvement in outcomes compared to those who did not experience improvement. Participants will include up to 40 patients who were treated with Brief CBT-CP. Participants will be interviewed about key components of the treatment and their perception of effectiveness. Interview data will be compared to the results of statistical analysis to help understand the mechanisms by which Brief CBT-CP is effective or identify areas for improvement. Results of this study will provide information needed to determine if Brief CBT-CP should be widely disseminated across VA primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age >=18 and <=79 years
* Conversant in English
* A diagnosis of musculoskeletal pain of >three months
* PEG score of >= 4 on pain intensity item and both interference items at screening
* BPI interference and pain intensity score of at least 4.0 at baseline
* If currently prescribed pain medication (other than topicals or NSAIDS), a stable dose in the last two months
* If currently prescribed psychiatric medicine, a stable dose in the last two months
* Established history of VA primary care utilization (i.e., at least one primary care visit in the past year)

Exclusion Criteria:

* Current or prior (past 12 months) engagement in psychotherapy or behavioral intervention provided by behavioral medicine services or specialty mental health for chronic pain.

  * Medication management through psychiatric services or an on-going course of mental health services for issues other than chronic pain are not excluded.
* Endorsement of imminent suicide risk
* Current significant substance use problems (i.e., alcohol, opioids, benzodiazepines, or other drugs)
* Unstable psychiatric status (e.g., active psychosis, current mania)
* Diagnosed with major or minor neurocognitive disorder
* Unwilling to have treatment sessions audio recorded
* Pending disability claim
* Recent or planned surgical/interventional procedure for pain

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P. Beehler, PhD, Principal Investigator — VA Western New York Healthcare System, Buffalo, NY
Locations (1):
- VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. The LDS will contain IPD that underlie results presented in publications.
Supporting Information: Study Protocol
Time Frame: IPD will be made available for up to three years starting six months after final publication.
Access Criteria: Data will be shared upon completion of a written request and within 90 days of a completed Data Use Agreement (DUA).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
Started | 92 | 92
Completed | 71 | 84
Not Completed | 21 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (13.4) | 57.8 (13.2) | 59.0 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 77 | 79 | 156
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 13 | 29
  White | 71 | 71 | 142
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12
Brief Pain Inventory -- Interference subscale (BPI-I) [Mean (Standard Deviation); unit: score on a measure] — This measure is a validated 7-item subscale that evaluates pain-related interference in daily activities and social and occupational functioning. Average scores range from 0 to 10, with higher scores indicating higher pain-related interference.
  score on a measure | 6.0 (1.5) | 6.1 (1.4) | 6.0 (1.5)
Brief Pain Inventory -- Pain Intensity subscale (BPI-P) [Mean (Standard Deviation); unit: score on a measure] — This measure is a validated 4-item subscale that evaluates pain intensity. Average scores range from 0 to 10, with higher scores indicating worse pain intensity.
  score on a measure | 5.5 (1.5) | 5.6 (1.4) | 5.6 (1.5)
Patient Health Questionnaire -- 9 (PHQ-9) [Mean (Standard Deviation); unit: score on a measure] — This 9-item measure of depressive symptoms is validated for use in primary care. Total scores range from 0 to 27, with higher scores indicating more depression symptoms.
  score on a measure | 8.0 (5.4) | 9.1 (6.2) | 8.5 (5.8)
World Health Organization Quality of Life - BREF (WHOQOL-BREF) to assess physical quality of life [Mean (Standard Deviation); unit: score on a measure] — This 26-item abbreviated version of the full-length WHOQOL measure evaluates quality of life in several domains such as social relationships and satisfaction with person-environment interactions. Scoring is by subscales representing four domains (i.e., physical health, psychological, social relationship, and environment). Transformed mean scores for each domain range from four to 20, with higher scores indicating greater quality of life in the respective domain.
  score on a measure | 11.7 (2.5) | 12.0 (2.9) | 11.9 (2.7)
World Health Organization Quality of Life - BREF (WHOQOL-BREF) to assess psychological health [Mean (Standard Deviation); unit: score on measure] — This 26-item abbreviated version of the full-length WHOQOL measure evaluates quality of life in several domains such as social relationships and satisfaction with person-environment interactions. Scoring is by subscales representing four domains (i.e., physical health, psychological, social relationship, and environment). Transformed mean scores for each domain range from four to 20, with higher scores indicating greater quality of life in the respective domain.
  score on measure | 14.8 (2.5) | 14.1 (2.9) | 14.5 (2.8)
World Health Organization Quality of Life - BREF (WHOQOL-BREF) to assess social quality of life [Mean (Standard Deviation); unit: score on a measure] — This 26-item abbreviated version of the full-length WHOQOL measure evaluates quality of life in several domains such as social relationships and satisfaction with person-environment interactions. Scoring is by subscales representing four domains (i.e., physical health, psychological, social relationship, and environment). Transformed mean scores for each domain range from four to 20, with higher scores indicating greater quality of life in the respective domain.
  score on a measure | 14.0 (2.7) | 14.0 (3.3) | 14.0 (3.0)
World Health Organization Quality of Life - BREF (WHOQOL-BREF) to assess environmental quality of li [Mean (Standard Deviation); unit: score on a measure] — This 26-item abbreviated version of the full-length WHOQOL measure evaluates quality of life in several domains such as social relationships and satisfaction with person-environment interactions. Scoring is by subscales representing four domains (i.e., physical health, psychological, social relationship, and environment). Transformed mean scores for each domain range from four to 20, with higher scores indicating greater quality of life in the respective domain.
  score on a measure | 15.9 (2.2) | 15.4 (2.4) | 15.7 (2.4)
Ability to Participate in Social Roles and Activities - short form (APSRA) [Mean (Standard Deviation); unit: Score on a measure] — This 8-item measure was developed to evaluate one's perceived ability to perform usual social roles and activities. Total scores range from eight to 40, with higher scores indicating better ability to participate in usual activities.
  Score on a measure | 27.0 (6.1) | 27.2 (5.9) | 27.1 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory -- Interference Subscale (BPI-I) to Assess Change at 12 Week Follow-up
Description: This measure is a validated 7-item subscale that evaluates pain-related interference in daily activities and social and occupational functioning. Average scores range from 0 to 10, with higher scores indicating higher pain-related interference.
Time Frame: 12-weeks
Measure: Mean (Standard Error); unit: score on instrument
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 71 | 84
score on instrument | 4.58 (.23) | 5.35 (.22)
Statistical Analysis 1: Comparison: Brief CBT for Chronic Pain and Treatment as Usual vs Treatment as Usual Only; Test type: Superiority; p = 0.026, Mixed Models Analysis; Mean Difference (Final Values) = 0.69, Standard Error of Mean 0.31

2. Secondary Outcome: Brief Pain Inventory -- Pain Intensity Subscale (BPI-P) to Assess Change at 12 Week Follow-up
Description: This measure is a validated 4-item subscale that evaluates pain intensity. Average scores range from 0 to 10, with higher scores indicating worse pain intensity.
Time Frame: 12-weeks
Measure: Mean (Standard Error); unit: score on intstrument
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 71 | 84
score on intstrument | 5.01 (0.18) | 5.43 (0.17)
Statistical Analysis 1: Comparison: Brief CBT for Chronic Pain and Treatment as Usual vs Treatment as Usual Only; Test type: Superiority; p = 0.124, Mixed Models Analysis — Adjusted for multiple comparisons; Mean Difference (Final Values) = 0.35, Standard Error of Mean 0.22

3. Secondary Outcome: Patient Health Questionnaire -- 9 (PHQ-9) to Assess Change at 12 Week Follow-up
Description: This 9-item measure of depressive symptoms is validated for use in primary care. Total scores range from 0 to 27, with higher scores indicating more depression symptoms.
Time Frame: 12-weeks
Measure: Mean (Standard Error); unit: score on instrument
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 71 | 84
score on instrument | 6.75 (0.57) | 8.10 (0.54)
Statistical Analysis 1: Comparison: Brief CBT for Chronic Pain and Treatment as Usual vs Treatment as Usual Only; Test type: Superiority; p = 0.746, Mixed Models Analysis — Adjusted for multiple comparisons; Mean Difference (Final Values) = 0.24, Standard Error of Mean 0.75

4. Secondary Outcome: World Health Organization Quality of Life - BREF (WHOQOL-BREF) to Assess Physical Health Change at 12 Week Follow up
Description: This 26-item abbreviated version of the full-length WHOQOL measure evaluates quality of life in several domains such as social relationships and satisfaction with person-environment interactions. Scoring is by subscales representing four domains (i.e., physical health, psychological, social relationship, and environment). Transformed mean scores for each domain range from four to 20, with higher scores indicating greater quality of life in the respective domain.
Time Frame: 12-weeks
Measure: Mean (Standard Error); unit: score on measure
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 71 | 84
score on measure | 13.016 (0.31) | 12.10 (0.29)
Statistical Analysis 1: Comparison: Brief CBT for Chronic Pain and Treatment as Usual vs Treatment as Usual Only; Test type: Superiority; p = 0.0002, Mixed Models Analysis — Adjusted for multiple comparisons; Mean Difference (Final Values) = -1.38, Standard Error of Mean 0.36

5. Secondary Outcome: World Health Organization Quality of Life - BREF (WHOQOL-BREF) to Assess Psychological Change at 12 Week Follow up
Description: as for outcome 4
Time Frame: 12-weeks
Measure: Mean (Standard Error); unit: score on a measure
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 71 | 84
score on a measure | 15.16 (0.31) | 13.85 (0.30)
Statistical Analysis 1: Comparison: Brief CBT for Chronic Pain and Treatment as Usual vs Treatment as Usual Only; Test type: Superiority; p = 0.046, Mixed Models Analysis — Adjusted for multiple comparisons; Mean Difference (Final Values) = -0.63, Standard Error of Mean 0.31

6. Secondary Outcome: World Health Organization Quality of Life - BREF (WHOQOL-BREF) to Assess Social Change at 12 Week Follow up
Description: as for outcome 4
Time Frame: 12-weeks
Measure: Mean (Standard Error); unit: score on a measure
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 71 | 84
score on a measure | 14.54 (0.37) | 13.85 (0.30)
Statistical Analysis 1: Comparison: Brief CBT for Chronic Pain and Treatment as Usual vs Treatment as Usual Only; Test type: Superiority; p = 0.161, Mixed Models Analysis — Adjusted for multiple comparisons; Mean Difference (Final Values) = -0.65, Standard Error of Mean 0.46

7. Secondary Outcome: World Health Organization Quality of Life - BREF (WHOQOL-BREF) to Assess Environmental Health Change at 12 Week Follow up
Description: as for outcome 4
Time Frame: 12-weeks
Measure: Mean (Standard Error); unit: score on a measure
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 71 | 84
score on a measure | 16.28 (0.25) | 15.67 (0.24)
Statistical Analysis 1: Comparison: Brief CBT for Chronic Pain and Treatment as Usual vs Treatment as Usual Only; Test type: Superiority; p = 0.719, Mixed Models Analysis — Adjusted for multiple comparisons; Mean Difference (Final Values) = -0.12, Standard Error of Mean 0.32

8. Secondary Outcome: Ability to Participate in Social Roles and Activities - Short Form (APSRA) to Assess Change at 12 Week Follow up
Description: This 8-item measure was developed to evaluate one's perceived ability to perform usual social roles and activities. Total scores range from eight to 40, with higher scores indicating better ability to participate in usual activities.
Time Frame: 12-weeks
Measure: Mean (Standard Error); unit: score on instrument
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 71 | 84
score on instrument | 28.32 (0.77) | 26.90 (0.73)
Statistical Analysis 1: Comparison: Brief CBT for Chronic Pain and Treatment as Usual vs Treatment as Usual Only; Test type: Superiority; p = 0.098, Mixed Models Analysis — Adjusted for multiple comparisons; Mean Difference (Final Values) = -1.61, Standard Error of Mean 0.97

ADVERSE EVENTS:
Time Frame: Enrollment to 12 week follow-up
Arm/Group | Brief CBT for Chronic Pain and Treatment as Usual | Treatment as Usual Only
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92
Serious Adverse Events (participants affected / at risk) | 2/92 | 4/92
Other Adverse Events (participants affected / at risk) | 12/92 | 10/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brief CBT for Chronic Pain and Treatment as Usual (N=92) | Treatment as Usual Only (N=92)
Evaluation for CVA (Vascular disorders) | 1 | 1
Rib fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Admitted for persistent cough and sore throat (Infections and infestations) | 0 | 1
Admitted for evaluation of syncope (Nervous system disorders) | 1 | 0
Admitted for abdominal pain (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brief CBT for Chronic Pain and Treatment as Usual (N=92) | Treatment as Usual Only (N=92)
Low back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Ankle pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Arm pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Elevated blood sugar (Metabolism and nutrition disorders) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 0
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1
Injuries due to assault (Injury, poisoning and procedural complications) | 1 | 0
Foot pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Abdominal pain and cramping (Gastrointestinal disorders) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 2
Cellulitus (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT04724694/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT04724694/ICF_000.pdf